CLINICAL TRIAL: NCT05506579
Title: Musculoskeletal Injuries, Pelvic Floor Dysfunctions and Menstrual Irregularities in Norwegian Rhythmic Gymnasts and Dancers - Observational and Cluster Randomized Controlled Studies
Brief Title: Prevention and Treatment of Injuries and Urinary Incontinence Among Norwegian Rhythmic Gymnasts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Responsible Party: Principal Investigator, Kari Bø, Professor, PhD, Physical therapist, Exercise scientist, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: MCDG2022
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Overuse Injury; Urinary Incontinence
Keywords: Overuse Injury; Urinary Incontinence; Rhythmic Gymnastics; Female athletes
MeSH Terms: conditions — Cumulative Trauma Disorders; Urinary Incontinence | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is an assessor blinded cluster randomized controlled trial with rhythmic gymnastics clubs as the unit of randomization. Two different interventions (preventive exercises for the knees, lower back and hip/groin and PFMT) for two different conditions (overuse injuries and UI) are combined in this design.
  After inclusion, all rhythmic gymnastics clubs will be randomly allocated 1:1 to preventive exercises for knee, lower back and hip/groin and PFMT or a control group with no intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Exercises for knees, lower back and hip/groin in an expanded warm up program. In addition, the warm up program will include pelvic floor muscle training (PFMT). The warm up program will in total take approximately 12-15 minutes to conduct each training.
  Interventions: Other: Exercises for knees, lower back, hip/groin and pelvic floor muscles in an expanded warm up program
- Control group (No Intervention): No intervention.

INTERVENTIONS:
Other: Exercises for knees, lower back, hip/groin and pelvic floor muscles in an expanded warm up program — Rhythmic gymnastics clubs allocated to the intervention group will be visited by a physiotherapist (the PhD candidate), which will perform thorough teaching of coaches and gymnasts on how to perform the exercises in the expanded warm up program. During the same visit, before commencing PFMT, the gymnasts will have an individual session were a portable 2D ultrasound machine (GE Healthcare -Logiq e R7, GE>12L-RS - 5-13 MHz Wideband Linear Probe) will be used to teach and assess ability to perform a correct PFM contraction. The probe is placed suprapubically and provides concurrent visible biofeedback of the PFM contraction. Adherence to the intervention will be registered weekly by the coach in a training diary and asked for as an additional question in the monthly OSTRC-H2 sent to the gymnasts. Reminders will be sent by phone to the coaches every week. To assure proper execution and motivation, the PhD candidate will perform one extra visit midterm.
  Arms: Intervention group

SUMMARY:
Overuse injuries are common among competitive Norwegian rhythmic gymnasts with a mean weekly prevalence of 37% [95% CI: 36 - 39%] and incidence of 4.2 new overuse injuries [95% CI: 3.6 - 4.9] per gymnast per year (Gram, M., Clarsen, B., & Bø, K., 2021). The knees, lower back and hip/groin were the most common injury locations. It has been postulated that reduced physical capacity (e.g strength, flexibility, stability) in the knees, lower back and hip/groin can increase the risk of injuries in rhythmic gymnastics.

In addition, more than 30% of the Norwegian rhythmic gymnasts experience urinary incontinence (UI), and 70% reported that UI negatively affected sports performance (Gram, M., & Bø, K., 2020). Few of the rhythmic gymnasts had any knowledge about the pelvic floor.

Hence, this assessor blinded cluster randomized controlled trial aims to find out whether the implementation of exercises targeting reduced physical capacity and pelvic floor dysfunction can prevent/reduce the prevalence of overuse injuries and UI.

DETAILED DESCRIPTION:
BACKGROUND

Norwegian rhythmic gymnasts have high prevalence and incidence of overuse injuries. Previous research on risk factors related to injuries in rhythmic gymnastics (RG) has implied that high weekly training load, hypermobility, poor technic and inappropriate training load increase the risk of injuries. A prospective study also found that previous injury increased the risk of injuries substantially (Gram, M., Clarsen, B., & Bø, K., 2021). Hence, injury prevention interventions should start at an early age to avoid the first injury. In addition, since the aetiology and mechanisms of injuries are multifactorial, with a well described complex interaction of internal and external risk factors making a gymnast more or less prone to sustain an injury, there might be a need to assess some internal risk factors more thoroughly. The modifiable internal risk factor physical capacity, e.g. strength, flexibility, stability, might be of particular interest, since lack of physical capacity can be thought of as a potential underlying cause in all of the above-mentioned risk factors. In addition, it is well known how persistent lack of physical capacity relative to the requirements in a sport might lead to injuries. With knees, lower back and hip/groin as the most commonly reported injury locations, clinical assessment of strength, flexibility and stability in these locations has been conducted in a cross-sectional study before this randomized controlled trial (RCT). Reduced physical capacity revealed in the cross-sectional study will be targeted/brought forward in the exercise program in the RCT.

The most common types of pelvic floor dysfunctions (PFD) are urinary incontinence (UI), anal incontinence (AI) and pelvic organ prolapse (POP). UI has high prevalence among female athletes participating in sports including jumping and running (high impact). A prevalence of 80% was found in young, nulliparous high-level trampoline jumpers in Sweden (Eliasson et.al., 2008). The prevalence among Norwegian rhythmic gymnasts was >30%, while Thyssen et.al. found that 56% of female Danish artistic gymnasts and 43% of dancers reported UI. UI negatively affects sports performance, and symptoms at young age is a risk factor of future UI developing during pregnancy and after childbirth. Hence, interventions toward prevention and treatment is necessary. While strength training of the pelvic floor muscles has 1A level of evidence/recommendation to treat UI in the general female population, and has no known adverse effects, there is little knowledge of this among young female athletes and dancers. Search on PubMed revealed only one RCT assessing the effect of pelvic floor muscle training on UI in female athletes. Ferreira et.al. randomized 32 female volleyball players to 3 months of pelvic floor muscle training or control, and found statistically significant improvement in the exercise group in frequency of leakage and urine loss measured during physical activity(p< 0.001). Hence, there seem to be a potential for prevention and treatment also in athletes exposed to heavy load towards the pelvic floor.

AIMS

The aims of this RCT are to investigate if implementation of prophylactic exercises targeting reduced capacity and pelvic floor dysfunction can prevent/lower the prevalence of overuse injuries and UI among Norwegian rhythmic gymnasts.

STUDY DESIGN AND METHODS

All rhythmic gymnastics clubs that are members of the Norwegian Gymnastics Federation and have gymnasts fulfilling the inclusion criteria will be invited to participate. The clubs are then randomly allocated to either an exercise or control group. Randomization will be provided by a person not involved in assessments of outcome.

All gymnasts in both groups will answer the "Oslo Sports Trauma Research Center Questionnaire on Health Problems" (OSTRC-H2) at baseline (including a part with background questions) and once each month during the intervention period. In addition, the gymnasts will answer the "International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form" (ICIQ-UI-SF) before and after the intervention period. After the intervention, the intervention group will answer the Global rating of change (GRC), a numerical 11-point scale to assess self-experienced effect and progress related to overuse injuries and UI.

ELIGIBILITY:
Inclusion Criteria:

* All rhythmic gymnastics clubs that are members of the Norwegian Gymnastics Federation and have gymnasts fulfilling the inclusion criteria will be invited to participate.
* Female rhythmic gymnasts ≥12 years of age training ≥3 days per week

Exclusion Criteria:

* Female rhythmic gymnasts <12 years of age training <3 days per week

Min Age: 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Rhythmic gymnastics is a female sport in Norway. Hence, the study will only include female gymnasts.
Enrollment: 205 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction in prevalence of overuse injuries in the knees, lower back and hip/groin | The gymnasts in both groups will answer the OSTRC-H2 at baseline (October 2022) and one time each month throughout the intervention period (last registration in June 2023)
  The Oslo Sports Trauma Research Center Questionnaire on Health Problems (OSTRC-H2) is a valid questionnaire to assess prevalence and severity of injuries in different anatomical areas.
Reduction in prevalence and bother of UI | The gymnasts in both groups will answer the ICIQ-UI-SF one time at baseline (October 2022) and one time when the intervention period has ended (June 2023)
  The International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form (ICIQ-UI-SF) is a reliable and valid questionnaire assessing prevalence, amount of leakage, bother and type of UI.

SECONDARY OUTCOMES:
Self-experienced effect and progress related to overuse injuries in the knees, lower back and hip/groin | The gymnasts in the intervention group will answer the GRC on time when the intervention period has ended (June 2023)
  Assessed by Global rating of change (GRC), a numerical 11-point scale, which has shown good test-retest reliability (ICC = 0.9).
Self-experienced effect and progress related to UI | The gymnasts in the intervention group will answer the GRC one time when the intervention period has ended (June 2023)
  Assessed by Global rating of change (GRC), a numerical 11-point scale, which has shown good test-retest reliability (ICC = 0.9).

CONTACTS AND LOCATIONS:
Overall Officials: Kari Bø, PhD, Study Chair — Norwegian School of Sport Sciences
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gram MCD, Clarsen B, Bo K. Injuries and illnesses among competitive Norwegian rhythmic gymnasts during preseason: a prospective cohort study of prevalence, incidence and risk factors. Br J Sports Med. 2021 Feb;55(4):231-236. doi: 10.1136/bjsports-2020-102315. Epub 2020 Aug 31. PMID 32868315
- [Background] Gram MCD, Bo K. High level rhythmic gymnasts and urinary incontinence: Prevalence, risk factors, and influence on performance. Scand J Med Sci Sports. 2020 Jan;30(1):159-165. doi: 10.1111/sms.13548. Epub 2019 Sep 30. PMID 31484216
- [Background] van Mechelen W, Hlobil H, Kemper HC. Incidence, severity, aetiology and prevention of sports injuries. A review of concepts. Sports Med. 1992 Aug;14(2):82-99. doi: 10.2165/00007256-199214020-00002. PMID 1509229
- [Background] Bahr R, Krosshaug T. Understanding injury mechanisms: a key component of preventing injuries in sport. Br J Sports Med. 2005 Jun;39(6):324-9. doi: 10.1136/bjsm.2005.018341. PMID 15911600
- [Background] Clarsen B, Bahr R, Myklebust G, Andersson SH, Docking SI, Drew M, Finch CF, Fortington LV, Haroy J, Khan KM, Moreau B, Moore IS, Moller M, Nabhan D, Nielsen RO, Pasanen K, Schwellnus M, Soligard T, Verhagen E. Improved reporting of overuse injuries and health problems in sport: an update of the Oslo Sport Trauma Research Center questionnaires. Br J Sports Med. 2020 Apr;54(7):390-396. doi: 10.1136/bjsports-2019-101337. Epub 2020 Feb 14. PMID 32060142
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278
- [Background] Bo K, Nygaard IE. Is Physical Activity Good or Bad for the Female Pelvic Floor? A Narrative Review. Sports Med. 2020 Mar;50(3):471-484. doi: 10.1007/s40279-019-01243-1. PMID 31820378
- [Background] de Mattos Lourenco TR, Matsuoka PK, Baracat EC, Haddad JM. Urinary incontinence in female athletes: a systematic review. Int Urogynecol J. 2018 Dec;29(12):1757-1763. doi: 10.1007/s00192-018-3629-z. Epub 2018 Mar 19. PMID 29552736
- [Background] Teixeira RV, Colla C, Sbruzzi G, Mallmann A, Paiva LL. Prevalence of urinary incontinence in female athletes: a systematic review with meta-analysis. Int Urogynecol J. 2018 Dec;29(12):1717-1725. doi: 10.1007/s00192-018-3651-1. Epub 2018 Apr 13. PMID 29654349
- [Background] Eliasson K, Edner A, Mattsson E. Urinary incontinence in very young and mostly nulliparous women with a history of regular organised high-impact trampoline training: occurrence and risk factors. Int Urogynecol J Pelvic Floor Dysfunct. 2008 May;19(5):687-96. doi: 10.1007/s00192-007-0508-4. Epub 2008 Jan 26. PMID 18224267
- [Background] Thyssen HH, Clevin L, Olesen S, Lose G. Urinary incontinence in elite female athletes and dancers. Int Urogynecol J Pelvic Floor Dysfunct. 2002;13(1):15-7. doi: 10.1007/s001920200003. PMID 11999199
- [Background] Bo K, Sundgot-Borgen J. Are former female elite athletes more likely to experience urinary incontinence later in life than non-athletes? Scand J Med Sci Sports. 2010 Feb;20(1):100-4. doi: 10.1111/j.1600-0838.2008.00871.x. PMID 19000097
- [Background] Dumoulin C, Cacciari LP, Hay-Smith EJC. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005654. doi: 10.1002/14651858.CD005654.pub4. PMID 30288727
- [Background] Ferreira, S., Ferreira, M., Carvalhais, A., Santos, P. C., Rocha, P., & Brochado, G. (2014). Reeducation of pelvic floor muscles in volleyball athletes. Revista da Associação Médica Brasileira, 60, 428-433.
- [Background] Avery K, Donovan J, Peters TJ, Shaw C, Gotoh M, Abrams P. ICIQ: a brief and robust measure for evaluating the symptoms and impact of urinary incontinence. Neurourol Urodyn. 2004;23(4):322-30. doi: 10.1002/nau.20041. PMID 15227649
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Derived] Gram MCD, Fagerland MW, Bo K. Pelvic floor muscle training by competitive rhythmic gymnasts at regular training sessions did not reduce urinary incontinence: a cluster-randomised trial. J Physiother. 2025 Apr;71(2):117-124. doi: 10.1016/j.jphys.2025.03.006. Epub 2025 Apr 1. PMID 40175233
- [Derived] Gram MCD, Fagerland MW, Bo K. Efficacy of a Rhythmic Gymnastics-Specific Injury Prevention Program: An Assessor-Blinded Cluster-Randomized Controlled Trial. Scand J Med Sci Sports. 2025 Feb;35(2):e70022. doi: 10.1111/sms.70022. PMID 39891397

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT05506579/SAP_000.pdf